CLINICAL TRIAL: NCT01256658
Title: A Cluster Randomized, Single-centre, Controlled, Parallel,12-month Prospective Study and Additional 12-month Follow-up in Africa of Malaria Incidence in a Community Setting Following Systematic Treatment of P. Falciparum Asymptomatic Carriers With Artemether-lumefantrine (Coartem® / Coartem® Dispersible)
Brief Title: A Community Setting Study of Malaria After Systematic Treatment of Symptomatic Carriers of P. Falciparum With COA566 (Coartem®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566B2401; CCOA566B2401E1 (Other: Novartis)
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-11

CONDITIONS: Malaria
Keywords: P. falciparum; malaria; asymptomatic carriers; bed-nets; ITN-insecticide-treated net; idiopathic trigeminal neuralgia; RDT-Rapid diagnostic test
MeSH Terms: conditions — Malaria; Trigeminal Neuralgia | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants received COA566 treatment for asymptomatic carriage of P. falciparum and for symptomatic malaria episodes.
  Interventions: Drug: COA566
- Control (Experimental): Participants received COA566 treatment for symptomatic malaria episodes only.
  Interventions: Drug: COA566

INTERVENTIONS:
Drug: COA566 — COA566 tablets or dispersible tablets twice daily during 3 days; dosage according to body weight.
  Other Names: Artemether-lumefantrine

SUMMARY:
This study assessed the impact of the systematic detection by Rapid Diagnostic Test (RDT) and treatment of asymptomatic carriers of malaria parasites (P. falciparum) with COA566 on a number of clinical malaria cases in children less than 5 years of age and the improvement of hemoglobin levels in the overall population.

ELIGIBILITY:
Inclusion:

* Subjects who were diagnosed as Asymptomatic Carrier (AC) by Rapid Diagnostic Test (RDT).
* Subjects who were diagnosed with a Symptomatic malaria episode, RDT-confirmed (SMRC)

Exclusion:

* Body weight <5 kg.
* Hypersensitivity to artemether-lumefantrine or to any of the excipients of the tablets or dispersible tablets.
* Presence of severe malaria signs and symptoms
* First trimester of pregnancy.
* Family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to prolong the QTc interval such as history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
* Taking drugs that are known to influence cardiac function and to prolong QTc interval, such as class IA and III: neuroleptics, antidepressant agents, certain antibiotics including some agents of the following classes: macrolides, fluoroquinolones, imidazole and triazole antifungal agents, certain non-sedating antihistamines.
* Known disturbances of electrolyte balance, e.g. hypokalemia or hypomagnesemia.
* Taking drugs which may be metabolized by cytochrome enzyme CYP2D6

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14075 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Burkina Faso (3):
  - Centre National de Recherche et de Formation sur le Paludisme, Ouagadougou, Ouagadougou
  - Novartis Investigative site, Ouagadougou, Ouagadougou
  - Novartis Investigative Site, Burkina Faso

REFERENCES:
- [Background] Ogutu B, Tiono AB, Makanga M, Premji Z, Gbadoe AD, Ubben D, Marrast AC, Gaye O. Treatment of asymptomatic carriers with artemether-lumefantrine: an opportunity to reduce the burden of malaria? Malar J. 2010 Jan 22;9:30. doi: 10.1186/1475-2875-9-30. PMID 20096111
- [Derived] Tiono AB, Guelbeogo MW, Sagnon NF, Nebie I, Sirima SB, Mukhopadhyay A, Hamed K. Dynamics of malaria transmission and susceptibility to clinical malaria episodes following treatment of Plasmodium falciparum asymptomatic carriers: results of a cluster-randomized study of community-wide screening and treatment, and a parallel entomology study. BMC Infect Dis. 2013 Nov 12;13:535. doi: 10.1186/1471-2334-13-535. PMID 24215306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an 18 clusters randomized study (1 cluster = 1 village). 14,075 participants were recruited during Period 1 (treatment); of these, 12,226 participants continued onto Period 2 (1 year follow-up) to assess longer term impact of initial intervention on malaria episodes. Period 2 was stopped and all participants discontinued.
Pre-assignment Details: During period 1 clusters were randomized 1:1 to either the control or the intervention arm (9 clusters per arm). In the intervention arm subjects were screened for asymptomatic carriage of P. falciparum status and treated with COA566. In both arms, subjects were treated for symptomatic malaria episodes. During period 2 there was no study treatment.
Period: Period 1
Arm/Group | Intervention | Control
Started | 6817 | 7258
Completed | 5897 | 6510
Not Completed | 920 | 748
Not completed — Lost to Follow-up | 837 | 661
Not completed — Withdrawal by Subject | 35 | 43
Not completed — Death | 48 | 44
Period: Period 2 - Follow up Only - No Treatment
Arm/Group | Intervention | Control
Started | 5854 (43 participants who completed period 1 did not enroll to continue on period 2) | 6372 (138 participants who completed period 1 did not enroll to continue on period 2)
Lost to Follow up | 71 | 77
Death | 6 | 8
Study Termination | 5777 (43 participants who completed period 1 did not enroll to continue on period 2) | 6287 (138 participants who completed period 1 did not enroll to continue on period 2)
Completed | 0 | 0
Not Completed | 5854 | 6372

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 6817 | 7258 | 14075
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.02 (20.67) | 22.62 (20.31) | 22.82 (20.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3656 | 3816 | 7472
  Male | 3161 | 3442 | 6603

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Malaria Episode, RDT-confirmed, With Parasitemia ≥5000/μL (SMRC5000s) Per Person-year in Infants and Children (<5 Years) in Post Community Screening Campaign (CSC) at Month 12 (Per Cluster)
Description: Data is presented "per cluster". Number of Symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000s) per person-year in infants and children (<5 years) in post Community Screening Campaign (CSC) at month 12 was detected by Rapid Diagnostic Test (RDT) (using a blood sample from each participant) and later confirmed to have a parasite density ≥5000/uL by microscopy.
  Number of SMRC5000: sum of all SMRC5000 for all infants and children (<5 years) in post CSC.
  Person-year observed: sum of duration (in days) for all infants and children (<5 years) in post CSC present in study /365.25.
  Number of SMRC5000 per person-year = number of SMRC5000/person-year observed.
Time Frame: Month 12 of period 1
Population: The number of units represents the number of clusters that include all randomized infants and children (<5 years) for which CSCs 1, 2, and 3 were conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: SMRC5000 per person-year
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1255 | 1235
Number analyzed (number of units) | 9 | 9
SMRC5000 per person-year | 1.69 (0.436) | 1.60 (0.526)

2. Primary Outcome: Change in Hemoglobin Level (g/dL) in Asymptomatic Carriers >6 Months of Age (Per Cluster)
Description: Data is presented "per cluster". Change in hemoglobin levels from day 1 to day 28 was measured using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each asymptomatic carrier from Community Screening Campaign 1 (CSC1), > 6 months of age, at day 1 and at day 28.
Time Frame: Day 1 and day 28 of period 1
Population: The number of units represents the number of clusters that include all randomized, > 6 months of age participants for which CSC1 was conducted, data was available and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: g/dL
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3523 | 3207
Number analyzed (number of units) | 9 | 9
g/dL
  Day 1 (n = 2387, 2116) | 11.81 (0.329) | 12.06 (0.345)
  Day 28 (n = 1136, 1091) | 12.33 (0.318) | 11.86 (0.373)

3. Secondary Outcome: Microscopy-confirmed Gametocyte Carriers at Community Screening Campaign 4 (CSC4) (Per Cluster)
Description: Data is presented "per cluster". Microscopy confirmed gametocyte carriers at Community Screening Campaign 4(CSC4) were assessed via microscopy at month 12 of period 1. Blood films were histologically treated and examined microscopically.
Time Frame: Month 12 - period 1
Population: The number of units represents the number of clusters that include all randomized participants for which CSC4 was conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Error); unit: participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 297 | 113
Number analyzed (number of units) | 9 | 9
participants | 4.9 (0.41) | 5.1 (0.41)

4. Secondary Outcome: Microscopy Confirmed Asymptomatic Carriers of P. Falciparum at Community Screening Campaign 4 (CSC4) (Per Cluster)
Description: Data is presented "per cluster". Microscopy confirmation of asymptomatic carriers of P. falciparum at Community Screening Campaign 4 (CSC4) was conducted at month 12. Blood films were histologically treated and examined microscopically. When it was ascertained that P. falciparum was present, a count of the asexual forms against leukocytes was made using a tally counter.
Time Frame: Month 12 - period 1
Population: The number of units represents the number of clusters that include all randomized participants for which CSC4 was conducted, data was available, and census data was obtained as per protocol.
Measure: Mean (Standard Error); unit: participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2023 | 815
Number analyzed (number of units) | 9 | 9
participants | 34.6 (1.86) | 37.6 (1.86)

5. Secondary Outcome: Change in Hemoglobin Level (g/dL) From Community Screening Campaign 1(CSC1)/Day 1 to Community Screening Campaign 4 (CSC4)/Day 1 (Per Cluster)
Description: Data is presented "per cluster". Comparison of hemoglobin level (g/dL) from Community Screening Campaign 1 (CSC1)/Day 1 to Community Screening Campaign 4 (CSC4)/Day 1 in infants and children (>6 months and <5 years) by study arm was measured using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each participant.
Time Frame: Day 1 (CSC1/day 1) and month 12 (CSC4/day 1) - period 1
Population: The number of units represents the number of clusters that include all infants and children (>6 months and <5 years) randomized participants for which CSCs 1 and 4 were conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: g/dL
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1167 | 1148
Number analyzed (number of units) | 9 | 9
g/dL
  CSC1/Day 1 (n= 819, 827) | 10.24 (0.371) | 10.04 (0.476)
  CSC4/Day 1 (n= 348,321) | 10.99 (0.267) | 11.13 (0.360)

6. Secondary Outcome: Number of Symptomatic Malaria Episode, RDT-confirmed, With Parasitemia ≥5000/μL (SMRC5000s) Per Person-year in Post Community Screening Campaign (CSC)
Description: Number of Symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000s) per person-year in post Community Screening Campaign (CSC), by study arm (individual level data) was detected by Rapid Diagnostic Test (RDT) (using a blood sample from each participant) and later confirmed to have a parasite density ≥5000/uL by microscopy.
  Number of SMRC5000: sum of all SMRC5000 for all subjects in post CSC. Person-year observed: sum of duration (in days) in post CSC for all subjects present in study /365.25.
  Number of SMRC5000 per person-year = number of SMRC5000/person-year observed.
Time Frame: 12 months - period 1
Population: Individual subject data from eligible clusters set defined as all randomized participants for which CSCs 1, 2, 3 and 4 were conducted, data was available, and census data were obtained as per protocol.
Measure: Number; unit: SMRC5000 per person-year
Arm/Group | Intervention | Control
Number analyzed (Participants) | 6817 | 7258
SMRC5000 per person-year | 0.45 | 0.39

7. Secondary Outcome: Number of Participants With Hospitalizations, Severe Malaria Episodes or Death Post Community Screening Campaign (CSC)
Description: Total number of participants (all ages) with hospitalizations, severe malaria episodes or death after Community Screening Campaign (CSC) was assessed.
Time Frame: 12 months - period 1
Population: Safety analyzable asymptomatic carriers set consisted of all consenting inhabitants from intervention clusters confirmed positive by RDT for P. falciparum asexual forms at any CSC or when migrating into the cluster, in the absence of clinical signs and symptoms who received at least one dose of COA566 to treat the diagnosed asymptomatic infection.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 6817 | 7258
participants
  Hospitalizations | 68 | 57
  Severe malaria episodes | 10 | 9
  Death | 31 | 31

8. Secondary Outcome: Number of Participants (Infants and Children (> 6 Months and < 5 Years)) With Hospitalizations, Severe Malaria Episodes or Death Post Community Screening Campaign (CSC)
Description: Total number of participants (infants and children (> 6 months and < 5 years)) with hospitalizations, severe malaria episodes or death after Community Screening Campaign (CSC) was assessed.
Time Frame: 12 months - period 1
Population: Safety analyzable carriers set consisted of all infants and children (> 6 months and < 5 years)) from intervention clusters confirmed positive for P. falciparum asexual forms at any CSC or when migrating into the cluster, who in the absence of clinical signs and symptoms received at least one dose of COA566 for the diagnosed asymptomatic infection.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1023 | 1040
participants
  Hospitalizations | 20 | 21
  Severe malaria episodes | 4 | 5
  Death | 2 | 2

9. Secondary Outcome: Mean of Microscopy-confirmed Asymptomatic Carriers From Community Screening Campaigns 1, 2, 3 and 4 (CSC1, CSC2, CSC3 and CSC4) (Per Cluster)
Description: Data is presented "per cluster". Mean number of asymptomatic carriers from Community Screening Campaigns 1, 2, 3 and 4 (CSC1, CSC2, CSC3 and CSC4) was measured by confirmed positive microscopy for P. falciparum asexual forms in participants with absence of clinical signs and symptoms of malaria.
  Mean measured in this analysis is the mean percent indicting the mean of percentages of cluster frequencies under the study arm for that particular category.
Time Frame: 12 months - period 1
Population: The number of units represents the number of clusters that include all randomized participants for which CSC 1, 2 3 and 4 was conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4859 | 3542
Number analyzed (number of units) | 9 | 9
participants
  CSC1/ day 1 (n= 2428, 1153) | 42.8 (5.67) | 47.5 (8.05)
  CSC2/ day 1 (n= 237, 833) | 4.1 (1.62) | 35.7 (4.94)
  CSC3/ day 1 (n= 171, 741) | 2.8 (0.92) | 32.2 (9.26)
  CSC4/ day 1 (n= 2023, 815) | 34.4 (3.92) | 37.8 (6.37)

10. Secondary Outcome: Mean Number of Microscopy-confirmed Gametocyte Carriers at Day 1 of Community Screening Campaign 1,2,3,4 (CSC1, CSC2, CSC3 and CSC4) (Per Cluster)
Description: Data is presented "per cluster". Mean number of gametocyte carriers at Day 1 for Community Screening Campaign 1,2,3,4 (CSC1, CSC2, CSC3 and CSC4) was measured using gametocyte assessments (prevalence and density) via microscopy.
  Mean measured in this analysis is the mean percent indicating the mean of percentages of cluster frequencies under the study arm for that particular category.
Time Frame: 12 months - period 1
Population: Eligible clusters set consisted of all randomized participants for which CSCs 1, 2, 3 and 4 were conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 878 | 633
Number analyzed (number of units) | 9 | 9
participants
  CSC1/Day 1 (n= 543, 246) | 9.5 (2.95) | 10.2 (4.54)
  CSC2/Day 1 (n= 33, 130) | 0.6 (0.38) | 5.5 (2.54)
  CSC3/Day 1 (n= 23, 144) | 0.4 (0.40) | 5.8 (1.77)
  CSC4/Day 1 (n= 279, 113) | 4.8 (1.34) | 5.1 (1.38)

11. Secondary Outcome: Number of Microscopy and qRT-PCR-confirmed Gametocyte Carriers at Community Screening Campaign 4 (CSC4)
Description: Number of gametocyte carriers at Community Screening Campaign 4 (CSC4) was measured via microscopy and confirmed using Quantitative Reverse Transcription PCR (qRT-PCR) at day 1 of CSC4.
Time Frame: Month 12 (CSC4/day 1) - period 1
Population: Individual subject data from eligible clusters set defined as all randomized participants for which CSC4 was conducted, data was available, and census data was obtained as per protocol.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1023 | 976
participants
  Positive | 508 | 462
  Negative | 514 | 511
  Not evaluable | 1 | 3

12. Secondary Outcome: Change in Hemoglobin Level (g/dL) From Community Screening Campaign 1 (CSC1)/Day 1 to CSC1/Day 28 in Infants and Children (>6 Months and <5 Years) for Asymptomatic Carriers at CSC1
Description: Change in hemoglobin level (g/dL) from Community Screening Campaign 1 (CSC1)/Day 1 to CSC1/Day 28 in infants and children (>6 Months and <5 Years) for asymptomatic carriers at CSC1 was measured via hemoglobin levels using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each participant. The anemic status is defined as follows: hemoglobin (Hb) <5 g/dL = severe anemia, Hb 5 to <8 g/dL = moderate anemia, Hb 8 to <11 g/dL = mild anemia, Hb ≥11 g/dL = no anemia).
Time Frame: Day 1 and day 28 - period 1
Population: Individual subject data from eligible clusters set defined as all infants and children (>6 months and <5 years) randomized for which CSC1 was conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Intervention | Control
Number analyzed (Participants) | 432 | 179
g/dL
  CSC1/Day 1 (n=432 ; 179 ) | 9.78 (1.763) | 9.67 (1.707)
  CSC1/Day 28 (n=406 ; 174 ) | 10.95 (1.543) | 10.17 (1.748)

13. Secondary Outcome: Anemia Status Based on Community Screening Campaign 1 (CSC1)/Day 1 in Infants and Children (>6 Months and <5 Years)
Description: Anemia status based on Community Screening Campaign 1 (CSC1)/Day 1 in infants and children (>6 months and <5 years) was measured via hemoglobin levels using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each participant. The anemic status is defined as follows: hemoglobin (Hb) <5 g/dL = severe anemia, Hb 5 to <8 g/dL = moderate anemia, Hb 8 to <11 g/dL = mild anemia, Hb ≥11 g/dL = no anemia).
Time Frame: Day 1 (CSC1/day 1) - period 1
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 819 | 348
participants
  CSC1/Day 1 Severe | 3 | 1
  CSC1/Day 1 Moderate | 80 | 36
  CSC1/Day 1 Mild | 458 | 195
  CSC1/Day 1 No symptoms | 278 | 116

14. Secondary Outcome: Anemia Status Based on Community Screening Campaign 4 (CSC4)/Day 1 in Infants and Children (>6 Months and <5 Years)
Description: Anemia status based on Community Screening Campaign 4 (CSC4/Day 1) in infants and children (>6 months and <5 years) was measured via hemoglobin levels using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each participant. The anemic status is defined as follows: hemoglobin (Hb) <5 g/dL = severe anemia, Hb 5 to <8 g/dL = moderate anemia, Hb 8 to <11 g/dL = mild anemia, Hb ≥11 g/dL = no anemia).
Time Frame: Month 12 (CSC4/day 1) - period 1
Population: Individual subject data from eligible clusters set defined as all infants and children (>6 months and <5 years) randomized for which CSC4 was conducted, data was available, and census data was obtained as per protocol.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 827 | 321
participants
  CSC4/Day 1 Severe | 1 | 1
  CSC4/Day 1 Moderate | 29 | 9
  CSC4/Day 1 Mild | 349 | 117
  CSC4/Day 1 No | 448 | 194

15. Secondary Outcome: Hemoglobin Level (g/dL) in Community Screening Campaign 1 (CSC1)/Day 1 and CSC4/Day 1 by Study Arm and Age Group (Per Cluster)
Description: Data is presented "per cluster". Hemoglobin levels at Community Screening Campaign 1 and 4 (CSC1 and CSC4) on day 1 per age group (5-9 years, 10-14 years, and ≥15 years) in the intervention versus the control arm was measured using the HemoCue® rapid test. This test was performed using a drop of blood collected from the fingertip of each participant.
Time Frame: Day 1 (CSC1/day 1) and month 12 (CSC4/day 1) - period 1
Population: The number of units represents the number of clusters that include all randomized participants (ages 5-9 years, 10-14 years, and ≥15 years) clusters for which CSC1 and CSC4 was conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: g/dL
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4677 | 2090
Number analyzed (number of units) | 9 | 9
g/dL
  CSC1 5- 9 years (n= 899, 431) | 11.63 (0.223) | 11.59 (0.239)
  CSC4 5 - 9 years (n= 900, 396) | 11.97 (0.224) | 12.13 (0.324)
  CSC1 10 - 14 years (n= 873, 380) | 12.32 (0.227) | 12.71 (0.301)
  CSC4 10 - 14 years (n= 837, 359) | 12.58 (0.161) | 12.72 (0.487)
  CSC1 >= 15 years (n= 2904, 1279) | 13.13 (0.304) | 13.49 (0.355)
  CSC4 >= 15 years (n= 2760, 1136) | 13.25 (0.167) | 13.42 (0.266)

16. Secondary Outcome: Percentage of COA566-treated Microscopy-confirmed Asymptomatic Carriers at Community Screening Campaign 1, 2 and 3 (CSC1, CSC2 and CSC3) With Parasitological Cure Rate at Day 7
Description: Percentage of participants with parasitological cure confirmed via microscopy at day 7 after treatment with COA566. This assessment was done on asymptomatic carriers from Community Screening Campaigns 1, 2 and 3 (CSC1, CSC2 and CSC3) from the intervention group only.
Time Frame: Day 7 of CSC1, CSC2 and CSC3 - period 1
Population: Treated asymptomatic carriers from CSC1, CSC2 and CSC3 confirmed by microscopy and treated with study medication. Subjects are counted multiple times if diagnosed and treated more than once during the study. Subjects missing day 7 parasitemia data are excluded. Percentages are based on the number of subjects treated with any formulation.
Measure: Number; unit: percentage of participants
Groups:
- Control: Not applicable to this outcome measure
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2450 | 0
percentage of participants
  CSC1 (n= 2151) | 99.5 |
  CSC2 (n=182) | 100 |
  CSC3 (n=117) | 96.7 |

17. Secondary Outcome: Percentage of Microscopy-confirmed Gametocyte Carriers Treated With COA566 for Asymptomatic Carriers
Description: Percentage of microscopy-confirmed gametocyte asymptomatic carriers treated with COA566 for asymptomatic carriers in Community Screening Campaign 1, 2 and 3 (CSC1, CSC2 and CSC3).
Time Frame: Day 1, day 7 and day 28 - period 1
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3970 | 0
percentage of participants
  CSC1 Day 1 (n= 3045) | 15.7 |
  CSC 1 Day 7 (n= 3045) | 1.4 |
  CSC 1 Day 28 (n= 3045) | 0.1 |
  CSC2 Day 1 (n= 850) | 2.6 |
  CSC2 Day 7 (n= 850) | 0.1 |
  CSC3 Day 1 (n= 75) | 4.0 |
  CSC3 Day 7 (n= 75) | 0 |

18. Secondary Outcome: Number of Asymptomatic Carriers With Increase in Hemoglobin Levels by at Least 0.5 g/dL From Community Screening Campaign 1 (CSC1) Infants and Children (>6 Months and <5 Years)- Individual Data
Description: Individual data of number of asymptomatic carriers with increase in hemoglobin levels by at least 0.5 g/dL from Day 1 to Day 28 from Community Screening Campaign 1 (CSC1) infants and children (>6 months and <5 years). Hemoglobin levels were measured using the HemoCue® rapid test. This test was performed with a drop of blood collected from the fingertip at Day 1 and at Day 28.
Time Frame: Day 1 to Day 28- period 1
Population: Individual subject data from eligible clusters set defined as all infants and children (>6 months and <5 years) randomized for which CSC1 was conducted, data was available, and census data was obtained as per protocol.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 434 | 180
participants | 288 | 79

19. Secondary Outcome: Number of Asymptomatic Carriers With Increase in Hemoglobin Levels by at Least 0.5 g/dL From Day 1 to Day 28 of Community Screening Campaign 1 (CSC1) in Infants and Children (>6 Months and <5 Years)- Cluster Data
Description: Data is presented "per cluster". Cluster data of number of asymptomatic carriers with increase in hemoglobin levels by at least 0.5 g/dL from Day 1 to Day 28 of Community Screening Campaign 1 (CSC1) in infants and children (>6 months and <5 years) was measured by Hemoglobin levels based on microscopy reading.
  Mean and Standard Deviation (SD) percent were measured indicating the mean and SD of percentages of cluster frequencies under the study arm for that particular category.
Time Frame: Day 1 to day 28 - period 1
Population: The number of units represents the number of clusters that include all infants and children (>6 months and <5 years) randomized for which CSC1 was conducted, data was available, and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 434 | 180
Number analyzed (number of units) | 9 | 9
participants | 66.1 (9.17) | 43.2 (12.45)

20. Secondary Outcome: Number of Symptomatic Malaria Episode, RDT-confirmed, With Parasitemia ≥5000/μL (SMRC5000) in Asymptomatic Carriers at Any Time of Diagnosis (Per Cluster)
Description: Data is presented "per cluster". Number of Symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000) in asymptomatic carriers by study arm from all inhabitants diagnosed at any time for asymptomatic carriers. Number of SMRC5000s is measured by Rapid diagnostic test (RDT) and later confirmed to have a parasite density ≥ 5000/uL by microscopy.
Time Frame: 12 months - period 1
Population: The number of units represents the number of clusters that include all participants randomized for which data on Symptomatic malaria episode, RDT-confirmed (SMRCs) were collected and census data were obtained as per protocol.
Measure: Mean (Standard Deviation); unit: percentage of participants
Units Other Than Participants: number of units
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2740 | 1381
Number analyzed (number of units) | 9 | 9
percentage of participants
  1 SMRC5000 | 15.25 (3.531) | 9.49 (3.123)
  2 SMRC5000 | 3.56 (1.258) | 2.78 (1.759)
  3 SMRC5000 | 1.28 (0.693) | 0.97 (0.934)
  >3 SMRC5000 | 0.67 (0.664) | 0.31 (0.417)

21. Secondary Outcome: Number of Asymptomatic Carriers With Complicated and Uncomplicated Episodes Combined
Description: Number of asymptomatic carriers diagnosed with 1 Symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000), 2 SMRC5000, 3 SMRC5000 and >3 SMRC5000 (complicated and uncomplicated episodes combined). Number of SMRC5000s is measured by Rapid diagnostic test (RDT) and later confirmed to have a parasite density ≥ 5000/uL by microscopy.
Time Frame: 12 months - period 1
Population: Individual subject data from eligible clusters set defined as all participants randomized for which data on Symptomatic malaria episode, RDT-confirmed (SMRCs) was collected and census data was obtained as per protocol.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2740 | 1381
participants
  1 SMRC5000 | 413 | 136
  2 SMRC5000 | 96 | 38
  3 SMRC5000 | 34 | 12
  >3 SMRC5000 | 17 | 5

22. Secondary Outcome: Cumulative Number of Subjects With Symptomatic Malaria Episode, RDT-confirmed, With Parasitemia ≥5000/μL From Week 1 to Week 50
Description: Cumulative number of asymptomatic carriers having Symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000) from Week 1 to Week 50, was measured from group of participants diagnosed as asymptomatic carriers at Community Screening Campaign (CSC1)/Day1. Number of participants affected before and after diagnosed with ≥1 symptomatic malaria episode, RDT-confirmed, with parasitemia ≥5000/μL (SMRC5000) (complicated and uncomplicated episodes combined). Number of SMRC5000s was detected by Rapid Diagnostic Test (RDT) using a blood sample from each participant and later confirmed to have a parasite density > or = 5000/uL by microscopy.
  Week (1-2) indicates day1 to day14, week (3-4) indicates day 15 to day 28, week (5-6) indicates day 29 to day 42, etc. After first diagnosis of asymptomatic carriers at CSC1/Day1.
Time Frame: Week 1 to Week 50
Population: Individual subject data from eligible randomized participants from Community Screening Campaign 1 (CSC1) for which data on Symptomatic malaria episode, RDT-confirmed (SMRCs) was collected and available form analysis and census data was obtained as per protocol.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2397 | 1138
participants
  Week (1-2) n at risk= 2397, 1138 | 1 | 4
  Week (3-4) n at risk= 2396, 1133 | 3 | 8
  Week (5-6) n at risk= 2391, 1129 | 4 | 12
  Week (7-8) n at risk= 2390, 1124 | 4 | 13
  Week (9-10) n at risk= 2390, 1123 | 4 | 15
  Week (11-12) n at risk= 2390, 1121 | 4 | 17
  Week (13-14) n at risk= 2390, 1103 | 4 | 18
  Week (15-16) n at risk= 2390, 1102 | 4 | 18
  Week (17-18) n at risk= 2390, 1102 | 4 | 18
  Week (19-20) n at risk= 2390, 1102 | 7 | 20
  Week (21-22) n at risk= 2337, 1083 | 30 | 24
  Week (23-24) n at risk= 2311, 1077 | 92 | 38
  Week (25-26) n at risk= 2246, 1063 | 188 | 59
  Week (27-28) n at risk= 2148, 1041 | 287 | 79
  Week (29-30) n at risk= 2047, 1020 | 347 | 98
  Week (31-32) n at risk= 1979, 996 | 391 | 114
  Week (33-34) n at risk= 1931, 979 | 421 | 121
  Week (35-36) n at risk= 1894, 968 | 440 | 130
  Week (37-38) n at risk= 1868, 956 | 460 | 144
  Week (39-40) n at risk= 1837, 935 | 477 | 149
  Week (41-42) n at risk= 1816, 927 | 483 | 154
  Week (43-44) n at risk= 1805, 920 | 486 | 158
  Week (45-46) n at risk= 1785, 913 | 490 | 159
  Week (47-48) n at risk= 1773, 910 | 492 | 161
  Week (49-50) n at risk= 1758, 904 | 493 | 161

ADVERSE EVENTS:
Time Frame: Safety assessed throughout duration of study.
Description: Safety assessments consisted of adverse events (AEs) and serious adverse events (SAEs) collection. AEs were collected during a period of 7 days from treatment administration start, for Asymptomatic Carriers and SMRCs only. SAEs were collected in both arms for the entire course of the study; hence the numbers in denominators are not consistent.
Groups:
- Intervention - Period 1: Participants received COA566 treatment for asymptomatic carriage of P. falciparum and for symptomatic malaria episodes.
- Control - Period 1: Participants received COA566 treatment for symptomatic malaria episodes only.
- Intervention - Period 2 - Follow-up Only: Participants from the intervention group of period 1 were followed up to assess longer term impact of initial intervention on malaria episodes. No treatment was given to participants during period 2.
- Control - Period 2- Follow-up Only: Participants from the control group of period 1 were followed up to assess longer term impact of initial intervention on malaria episodes. No treatment was given to participants during period 2.
Arm/Group | Intervention - Period 1 | Control - Period 1 | Intervention - Period 2 - Follow-up Only | Control - Period 2- Follow-up Only
Serious Adverse Events (participants affected / at risk) | 156/4826 | 134/2275 | 23/467 | 39/386
Other Adverse Events (participants affected / at risk) | 0/4826 | 0/2275 | 0/467 | 0/386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention - Period 1 (N=4826) | Control - Period 1 (N=2275) | Intervention - Period 2 - Follow-up Only (N=467) | Control - Period 2- Follow-up Only (N=386)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2
CARDIAC FAILURE (Cardiac disorders) | 2 | 1 | 0 | 1
HEART DISEASE CONGENITAL (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
SICKLE CELL ANAEMIA (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
SICKLE CELL ANAEMIA WITH CRISIS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
CONJUNCTIVAL PALLOR (Eye disorders) | 0 | 0 | 1 | 0
EYELID OEDEMA (Eye disorders) | 0 | 1 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 4 | 0 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1 | 1 | 2
FOOD POISONING (Gastrointestinal disorders) | 3 | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1 | 0 | 0
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 2 | 0 | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
LIP OEDEMA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 14 | 16 | 1 | 1
ASTHENIA (General disorders) | 0 | 1 | 0 | 1
DEATH (General disorders) | 11 | 13 | 2 | 1
PYREXIA (General disorders) | 5 | 4 | 3 | 0
SUDDEN DEATH (General disorders) | 2 | 1 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 4 | 1 | 0 | 1
BREAST ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 3 | 2 | 0 | 1
EXTRAPULMONARY TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 7 | 5 | 1 | 0
GASTROENTERITIS SHIGELLA (Infections and infestations) | 0 | 0 | 0 | 1
HEPATIC AMOEBIASIS (Infections and infestations) | 0 | 0 | 0 | 1
HIV INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
HYDROCELE MALE INFECTED (Infections and infestations) | 0 | 0 | 1 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0 | 1
INFECTION PARASITIC (Infections and infestations) | 0 | 1 | 2 | 0
MALARIA (Infections and infestations) | 42 | 39 | 9 | 8
MENINGITIS (Infections and infestations) | 1 | 4 | 0 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0
ORCHITIS (Infections and infestations) | 1 | 0 | 0 | 1
PARASITIC GASTROENTERITIS (Infections and infestations) | 1 | 2 | 0 | 0
PERITONEAL TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 28 | 23 | 3 | 7
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1 | 0 | 1
SEPSIS (Infections and infestations) | 1 | 2 | 0 | 1
TUBERCULOSIS (Infections and infestations) | 0 | 1 | 0 | 0
TYPHOID FEVER (Infections and infestations) | 2 | 6 | 1 | 1
CHEMICAL POISONING (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
SNAKE BITE (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
COMA (Nervous system disorders) | 0 | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 2 | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 1 | 0
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2 | 3 | 1 | 2
ABORTION THREATENED (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 1
CERVIX DYSTOCIA (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
COMPLICATION OF DELIVERY (Pregnancy, puerperium and perinatal conditions) | 3 | 2 | 1 | 1
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0
FOETAL MALPRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
POLYHYDRAMNIOS (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0
THIRD STAGE POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
UTERINE CERVICAL LACERATION DURING LABOUR (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
AFFECTIVE DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 2 | 0 | 0 | 0
PERSONALITY CHANGE (Psychiatric disorders) | 0 | 1 | 0 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 2 | 3 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 4 | 3 | 0 | 0
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 1 | 0 | 0
EPIDIDYMITIS (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
TESTICULAR TORSION (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
ASTHMATIC CRISIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
BRONCHOPNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.